CLINICAL TRIAL: NCT06538792
Title: Effect of Proprioception and Muscle Strength on Kinesiophobia After Anterior Cruciate Ligament Reconstruction
Brief Title: Proprioception, Muscle Strength and Kinesiophobia After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Pysiotherapy and Rehabilitation Department, Bezmialem Vakif University
Other Study IDs: Ka24-2
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fear of re-injury after anterior cruciate ligament reconstruction surgery (ACLR) affects individuals' return to sports and physical activity negatively. The aim of this study is to evaluate the effects of proprioception and muscle strength on kinesiophobia in patients who have undergone anterior cruciate ligament reconstruction surgery.

DETAILED DESCRIPTION:
Factors such as graft type, patient age, activity level and athletic experience, as well as psychological factors such as psychological readiness for return to sports, fear of re-injury, and motivation during the rehabilitation process, affect returning to sports after ACLR. Fear is a psychological reaction that occurs after injury and is clearly seen during the period when athletes continue to actively participate in sports. Individuals' confidence in their knees and pain after surgery affect their fear of movement.

While kinesiophobia provides benefits in protecting injured body parts in the acute phase of pain, it can lead to inactivity, emotional stress and risk of re-injury in the long term. Kinesiophobia changes the biomechanics of movements and pain perception. Insufficient muscle strength and instability in the knee negatively affect confidence in the knee. The aim of this study is to evaluate the effects of proprioception and muscle strength on kinesiophobia in patients who have undergone anterior cruciate ligament reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35
* History of ACL reconstruction surgery at least 6 months ago

Exclusion Criteria:

* History of previous lower extremity surgery
* History of lower extremity injury within the last 6 months
* Having a vestibular or neurologic pathology that would affect balance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have undergone ACL reconstruction surgery will be recruited from the Department of the Orthopaedics and Traumatology, Bezmialem Vakıf University Hospital.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | Baseline
  The Tampa Kinesiophobia Scale consists of seventeen items. Scores obtained from the scale range from 17 to 68, with higher scores indicating greater severity of kinesiophobia.
Joint position sense | Baseline
  Measurement of knee joint position sense by the active and passive repositioning technique with isokinetic dynamometer at 30˚ and 60˚.The deviation from the target angle is recorded in degrees. A high deviation from the target angle indicates a deficiency in proprioceptive sense.
Muscle strength | Baseline
  Assessment for knee extensor and flexor muscles with isokinetic dynamometer at 60 º/sec and 240º/sec angular velocity. The peak torque value (Nm), which is measured by the device and indicates the maximum force the subject can reach, will be used in the assessment.
Dynamic stability | Baseline
  The single leg dynamic stability test by the Biodex Balance System® (Biodex Medical Systems, Inc. USA). Low values of the stability index indicate better balance and stability, while higher scores indicate a lower ability to maintain postural stability.

SECONDARY OUTCOMES:
Return to sports after ACL injury | Baseline
  The ACL Return to Sports after Injury (ACL-RSI) scale is a 12-item scale, scored from 0 to 10, that evaluates psychological readiness for return to sports after ACL injury. High scores indicate positive psychological readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Alpay, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)